CLINICAL TRIAL: NCT00943735
Title: A 13-Week, Single-Arm, Open-Label, Multicenter Study To Evaluate Refill Adherence And Satisfaction With Fesoterodine Plus "Your Way" Patient Support Plan In Patients With Symptoms Of Overactive Bladder.
Brief Title: This Is An Open-Label Study To Evaluate Fesoterodine Plus "Your Way" Patient Support Plan In Patients With Symptoms Of Overactive Bladder
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A0221078
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Results first posted 2012-03-15 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder Incontinence Adherence Behavioral interventions
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fesoterodine arm: subjects who present with OAB symptoms during medical office visits and who appear to be candidates for fesoterodine therapy
  Interventions: Drug: Fesoterodine; Behavioral: Your Way

INTERVENTIONS:
Drug: Fesoterodine — Fesoterodine 4 mg and 8 mg QD
Behavioral: Your Way — early intervention after treatment initiation and before patients have an opportunity to discontinue medication; reinforcing the treatable nature of OAB

SUMMARY:
The primary objective of the study is to assess the level of medication adherence observed among subjects receiving a specific combination of education and support materials (YourWay plan) along with a prescription for fesoterodine.

DETAILED DESCRIPTION:
This is a non-interventional, observational study. Study investigators will recruit symptomatic, fesoterodine-naïve subjects when they present with OAB symptoms during regularly-scheduled physician visits fesoterodine-naïve subjects with OAB symptoms present during regularly-scheduled physician visits

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients >=18 years old
* Eligible for receiving Toviaz 4mg or 8mg QD treatment based on the approved US label.

Exclusion Criteria:

* Female subjects who are pregnant, lactating, or who are intending to become pregnant within 28 days after the completion of the study (use of contraceptives is not required to participate in the study)
* Have participated in any other studies involving study drugs within 30 days prior to entry in the study
* Subjects who have previously taken fesoterodine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: fesoterodine-naïve subjects with OAB symptoms present during regularly-scheduled physician visits
Sampling Method: Non-Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221078

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, observational study. Study investigators contacted through prescription records in the IMS Longitudinal prescription (LRx) Database recruited symptomatic, fesoterodine-naive subjects (N=788 recruited; 774 entered) when they presented with overactive bladder (OAB) symptoms during regularly-scheduled physician visits.
Pre-assignment Details: The use and dosage recommendations for fesoterodine 4 milligram (mg) or 8 mg tablet taken by mouth (PO) once daily (QD) adhered completely to the approved product label and was adjusted solely according to medical and therapeutic necessity.
Groups:
- Fesoterodine 4 mg or 8 mg: Fesoterodine 4 mg or 8 mg tablet PO, QD
Period: Overall Study
Arm/Group | Fesoterodine 4 mg or 8 mg
Started | 774
Per Protocol Population | 500
Completed | 742
Not Completed | 32
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 8
Not completed — Death | 1
Not completed — Other | 8
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 774
Age, Customized [Number; unit: participants]
  18 to 24 years | 5
  25 to 44 years | 119
  45 to 64 years | 325
  ≥ 65 years | 325
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 593
  Male | 181

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Filled at Least 90 Days Supply of Fesoterodine (4mg QD or 8mg QD) Within 90 Days of Study Enrollment
Description: Prototypical pattern for meeting primary endpoint was to fill 3 separate prescriptions (Rx), each for a 30-day supply between enrollment and Day 90. Rx fills could happen as early as Day 0, 30, and 60 of the study period. Participants could also have chosen to wait until their 14-day medication sample was exhausted before receiving their first fill. Investigators received no prescribing restrictions, but were advised not to write Rx for a 90-day supply of fesoterodine at enrollment visit. Participants whose first observed Rx was for a ≥90-day supply were non-evaluable for the primary endpoint.
Time Frame: Enrollment (Day 0) up to 90 days
Population: Per Protocol (PP) population: all participants who returned a signed informed consent form (Intent to Treat) and enrollment questionnaire, had evidence of ≥1 prescription in LRx database for any medication class, and did not receive an initial fesoterodine prescription for ≥ a 90-day supply.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 500
percentage of participants | 10.4 [7.7 to 13.1]

2. Secondary Outcome: Percentage of Participants Who Filled at Least One Fesoterodine Prescription During the Study Period (Primary Adherence)
Description: The prototypical pattern was to fill 3 separate prescriptions, each for a 30-day supply, between the enrollment date and Day 90 of the study period; these prescription fills could happen as early as Day 0, 30, and 60 of the study period. Primary adherence was met if the participant filled at least 1 fesoterodine prescription during the study period.
Time Frame: Enrollment (Day 0) up to 90 days
Population: PP population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 500
percentage of participants | 26.2 [22.5 to 29.9]

3. Secondary Outcome: Percentage of Participants Who Filled at Least Two Fesoterodine Prescriptions (First Refill) During the Study Period
Description: The prototypical pattern was to fill 3 separate prescriptions, each for a 30-day supply, between the enrollment date and Day 90 of the study period; these prescription fills could happen as early as Day 0, 30, and 60 of the study period. At enrollment, the Investigator provided participants with a prescription for fesoterodine 4mg or 8mg to be filled at a pharmacy of their choice. The first refill indicated that 2 fesoterodine prescriptions had been filled.
Time Frame: Enrollment (Day 0) up to 90 days
Population: PP population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 500
percentage of participants | 13.4 [10.5 to 16.3]

4. Secondary Outcome: Percentage of Participants Who Visited the YourWay Website
Description: YourWay plan was available and accessible to all participants prescribed fesoterodine, but was not defined as an explicit or required component. Plan included motivational support for taking fesoterodine and behavioral interventions shown in clinical studies to improve participants' Overactive Bladder (OAB) outcomes. Objectives included intervening quickly after treatment initiation, before participants had an opportunity to discontinue medication, reinforcing the treatable nature of OAB, and setting appropriate expectations for onset of action with therapy and degree of symptom improvement.
Time Frame: Baseline up to 90 days
Population: PP population; N=CATI response valid N: Participants' interview responses were reported via a computer-assisted telephone interview (CATI) with a live interviewer on or around Day 86 of the study period. Participants may have omitted responses to individual items; valid N, therefore, may have varied from response to response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 337
percentage of participants | 28.8 [24.0 to 33.9]

5. Secondary Outcome: Among Participants Who Used the YourWay Website, the Percentage of Participants Who Agreed That the Website Was Useful
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 337
percentage of participants | 3.0 [1.4 to 5.4]

6. Secondary Outcome: Percentage of Participants Who Reported Having Read the YourWay Plan Materials Received From Their Physician or From the Resource Kit
Description: YourWay plan included a starter pack with a 14-day supply of 4 mg or 8 mg fesoterodine; guidebook for YourWay plan components and lifestyle modification tips; plan progress tracker with additional lifestyle tips; plan enrollment form. About 1 week after plan enrollment, participants received a resource kit by mail which included: a cover letter; brochures for "Core 4" elements (food and drink, teach your bladder, daily fesoterodine, and track your progress); bladder diary and "track your progress" brochure; and recipes using bladder-friendly foods.
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 335
percentage of participants | 97.3 [95.0 to 98.8]

7. Secondary Outcome: Percentage of Participants Who Reported Having Adopted Lifestyle Changes to Help Improve Their Overactive Bladder (OAB) Symptoms
Description: The use of the YourWay plan was optional but was available to all participants and included guidance for food and drink choices, bladder training, treatment compliance, and use of a daily tracker.
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 339
percentage of participants | 85.3 [81.0 to 88.9]

8. Secondary Outcome: Percentage of Participants Who Reported That They Made Bladder-friendly Food and Drink Choices
Description: The use of the YourWay plan was optional but was available to all participants and included bladder-friendly food and drink choices and recipes as well as information for maintaining hydration and avoidance of potential bladder irritants (such as caffeine, citrus fruits and juices, artificial sweeteners, tomato-based foods, soda, alcohol, and spicy foods).
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 336
percentage of participants | 82.4 [77.9 to 86.4]

9. Secondary Outcome: Percentage of Participants Who Reported That They Trained Their Bladder to "Wait"
Description: The use of the YourWay plan was optional but was available to all participants and included bladder training techniques such as to urinate each day when getting up and before going to bed, gradually increasing the amount of time between urinating, staying with timing goals whether there was a need to urinate or not, and bladder control tips (such as pelvic floor muscle squeeze, sit down and take 5 deep breaths, or stating "I'm the boss - not my bladder").
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 335
percentage of participants | 86.6 [82.4 to 90.0]

10. Secondary Outcome: Percentage of Participants Who Reported That They Took Toviaz® (Fesoterodine) as Directed
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 327
percentage of participants | 93.9 [90.7 to 96.2]

11. Secondary Outcome: Percentage of Participants Who Reported That They Recorded Their Treatment Goals in the Daily Core 4 Tracker
Description: YourWay Daily Core 4 Tracker to track daily progress in the 4 core areas of food and drink (make more informed choices), teach your bladder (train your bladder to "wait"), daily Toviaz® (always take as directed), and keep track (share with your doctor).
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 340
percentage of participants | 56.8 [51.7 to 61.9]

12. Secondary Outcome: Percentage of Participants Who Reported That They Kept Track of Symptoms in the 12 Week Tracker Bladder Diary
Description: For each week, the 12 Week Tracker included a participant determined weekly goal, a reminder to fill the prescription (if appropriate interval), participant reported progress in response to "this week I did well at", and a 7-day Daily Core 4 Tracker checklist (food and drink, teach your bladder, daily fesoterodine, and track your progress).
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 339
percentage of participants | 57.4 [52.4 to 62.4]

13. Secondary Outcome: Percentage of Participants Who Reported That They Let Their Doctor Know How They Were Doing With the YourWay Plan
Description: Participants were recruited for study participation when they presented with OAB symptoms during regularly-scheduled physician visits; screening and enrollment occurred during the same visit. Follow-up visits could be scheduled per standard clinical practice.
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 332
percentage of participants | 56.6 [51.4 to 61.7]

14. Secondary Outcome: Percentage of Participants Who Agreed That They Found the YourWay Program Materials Easy to Understand
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 335
percentage of participants | 91.9 [88.5 to 94.6]

15. Secondary Outcome: Percentage of Participants Who Agreed That the YourWay Program Provided a Good Amount of Information
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 334
percentage of participants | 95.5 [92.7 to 97.5]

16. Secondary Outcome: Percentage of Participants Who Agreed That the YourWay Plan Provided a Strong Support System That Participants Could Count on for Information and Advice
Description: YourWay participants received 6 telephone calls from an automated speech-recognition system over a period of approximately 11 weeks. The calls included reinforcement of treatment participation, treatment expectations, compliance, general health messages regarding OAB, review of training materials, optional weekly email communication, and a wrap-up call which included a summary of lessons learned from each of the Core 4 lessons calls and guidance to find additional information about medication and lifestyle tips to support management of OAB symptoms.
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 333
percentage of participants | 81.7 [77.1 to 85.7]

17. Secondary Outcome: Percentage of Participants Who Agreed That They Were Able to Incorporate the YourWay Plan Into Their Lives
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 332
percentage of participants | 81.6 [77.0 to 85.6]

18. Secondary Outcome: Percentage of Participants Who Agreed That the YourWay Plan Helped Them Play a More Active Role in Managing Their Condition
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 336
percentage of participants | 79.9 [75.8 to 84.1]

19. Secondary Outcome: Percentage of Participants Who Agreed That They Understood What to Expect From Their OAB Medication, Toviaz® (Fesoterodine)
Description: Product indication and safety information was provided to all participants by the investigator and / or within the YourWay plan program information.
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 331
percentage of participants | 88.2 [84.2 to 91.5]

20. Secondary Outcome: Percentage of Participants Who Agreed That They Learned Something About Their Condition
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 338
percentage of participants | 87.0 [82.9 to 90.4]

21. Secondary Outcome: Percentage of Participants Who Agreed That They Increased Their Knowledge of Healthy Bladder Behaviors
Description: The use of the YourWay plan was optional but was available to all participants and included healthy bladder behaviors such as setting and maintaining personal goals and choice of bladder-friendly food and drinks.
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 339
percentage of participants | 85.3 [81.0 to 88.9]

22. Secondary Outcome: Percentage of Participants Who Agreed That They Understand OAB is a Chronic Condition That Can be Successfully Managed, But Generally Not Cured
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 337
percentage of participants | 93.8 [90.6 to 96.1]

23. Secondary Outcome: Percentage of Participants Who Reported They Felt Confident That They Could Manage Their OAB as a Result of the YourWay Plan
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 330
percentage of participants | 72.4 [67.3 to 77.2]

24. Secondary Outcome: Percentage of Participants Who Reported They Were Satisfied With the Overall Content of the YourWay Plan
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 336
percentage of participants | 86.9 [83.3 to 90.4]

25. Secondary Outcome: Percentage of Participants Who Reported They Were Satisfied With the Participant Support Telephone Calls
Description: as for outcome 16
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 325
percentage of participants | 78.5 [73.6 to 82.8]

26. Secondary Outcome: Percentage of Participants Who Reported They Were Satisfied With the Treatment Goals and Bladder Symptoms Progress Trackers
Description: Treatment goals and bladder symptoms progress trackers were incorporated in the 12 Week Tracker which included a participant determined weekly goal, a reminder to fill the prescription (if appropriate interval), participant reported progress in response to "this week I did well at", and a 7-day Daily Core 4 Tracker checklist (food and drink, teach your bladder, daily fesoterodine, and track your progress).
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 328
percentage of participants | 74.1 [69.0 to 78.7]

27. Secondary Outcome: Percentage of Participants Who Reported They Were Satisfied With Their Physician
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 334
percentage of participants | 93.4 [90.2 to 95.8]

28. Secondary Outcome: Percentage of Participants Who Reported the YourWay Plan Encouraged Their Use of Toviaz® (Fesoterodine)
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 328
percentage of participants | 69.2 [63.9 to 74.2]

29. Secondary Outcome: Percentage of Participants Who Agreed That They Had a Good Understanding About Their Condition and How to Treat it
Time Frame: Baseline up to 90 days
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 335
percentage of participants | 89.6 [85.8 to 92.6]

30. Secondary Outcome: Comparison of Percentage of Participants Who Agreed That They Had a Good Understanding About Their Condition and How to Treat it, Between Enrollment Date and End of Study CATI Interview
Time Frame: Enrollment (Day 0) up to 90 days
Population: PP population; (n)=CATI response valid n at observation. Participants' interview responses were reported via a computer-assisted telephone interview (CATI) with a live interviewer on or around Day 86 of the study period. Participants may have omitted responses to individual items; valid n, therefore, may have varied from response to response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fesoterodine 4 mg or 8 mg
Number analyzed (Participants) | 500
percentage of participants
  Good understanding at enrollment (n=500) | 78.4 [75.5 to 81.3]
  Good understanding at end of study (n=335) | 89.6 [85.8 to 92.6]

ADVERSE EVENTS:
Time Frame: Enrollment (Day 0) up to 28 days after last dose of study treatment
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Fesoterodine 4 mg or 8 mg
Serious Adverse Events (participants affected / at risk) | 13/774
Other Adverse Events (participants affected / at risk) | 100/774
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 mg or 8 mg (N=774)
Arrhythmia (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Hypertensive heart disease (Cardiac disorders) | 1
Vision blurred (Eye disorders) | 1
Chest pain (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Activities of daily living impaired (Social circumstances) | 1
Colporrhaphy (Surgical and medical procedures) | 1
Transurethral bladder resection (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fesoterodine 4 mg or 8 mg (N=774)
Cataract (Eye disorders) | 1
Dry eye (Eye disorders) | 4
Vision blurred (Eye disorders) | 11
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 25
Diarrhoea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 22
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Oesophageal pain (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Cystitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Balance disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 8
Somnolence (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Mood swings (Psychiatric disorders) | 1
Nightmare (Psychiatric disorders) | 2
Bladder obstruction (Renal and urinary disorders) | 1
Cystitis interstitial (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 5
Micturition urgency (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 6
Urge incontinence (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 8
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.